CLINICAL TRIAL: NCT04248218
Title: Randomized Trial of Active Rehabilitation for Acute Pediatric Concussions
Brief Title: Concussion Active Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Jeremy Root, Assistant Professor of Pediatrics and Emergency Medicine, George Washington Univ School of Medicine, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro0012220
Record Dates: First submitted 2020-01-03; First posted 2020-01-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Pediatric ALL; Concussion, Mild; Concussion, Brain; Concussion, Intermediate
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Brain Concussion

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized control trial of pediatric patients in the emergency department (ED) diagnosed with an acute concussion.
  The randomization plan will include randomization based on sex.
  Group A: active care Group B: routine/standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal/Control (No Intervention): Control Group/Standard Care
- Active Rehabilitation Group/Case (Active Comparator): Active Rehabilitation Cohort/Intervention
  Interventions: Behavioral: Active Rehabilitation Group/Case

INTERVENTIONS:
Behavioral: Active Rehabilitation Group/Case — If the patient is in the active rehabilitation group, the patient will receive instructions based on the latest CDC concussion management guidelines that specify a symptom-limited progressive return to full activities. This group will be instructed to take at least 10,000 steps a day for five days on their pedometers. In addition, they will also watch a two-minute video by the PI and research team reinforcing the active rehabilitation instructions.
  Arms: Active Rehabilitation Group/Case

SUMMARY:
In this study, the investigator plans a randomized trial of active rehabilitation and standard care for acute concussion management. The investigator hypothesizes that patients with acute concussions managed with active rehabilitation will have decreased risk of prolonged concussion symptoms.

DETAILED DESCRIPTION:
Specific Aims:

To compare the risk of prolonged concussion symptoms (PCS) between an active rehabilitation and a standard care cohort after an acute concussion.

To determine if active rehabilitation compared to routine care reduces the risk of PCS for high-risk patients.

This is a prospective randomized control trial of pediatric patients in the emergency department (ED) diagnosed with an acute concussion. Patients 8-18 years old with an acute concussion diagnosis will be eligible. All patients will receive pedometers to monitor their activity levels. If the patient is in the control group the patient will receive standard concussion management per the treating ED physician. Patients in the active rehabilitation group will receive instructions based on the latest CDC concussion management guidelines that specify a symptom-limited progressive return to full activities. This group will be instructed to take at least 10,000 steps a day for five days on their pedometers.

One to five days after the ED concussion diagnosis a trained research coordinator will call all subjects to reinforce the management plan.

28 to 32 days post ED concussion diagnosis, research assistants will contact subjects via email or phone call to complete the concussion symptoms inventory.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with an acute concussion within 48 hours
* Patient greater than 8 and less than 19 years old

Exclusion Criteria:

* Major psychiatric diagnosis (bipolar disorder, major depression, does NOT include ADHD/ADD)
* Cognitive delay
* GCS < 14
* positive findings on head CT
* Any patient with intracranial surgery, pathology or instrumentation (e.g. VP shunt, brain tumor etc)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
We will measure and compare the relative risk of prolonged concussion symptoms (PCS) between an active rehabilitation and a standard care cohort one month after an acute concussion. | 28 to 32 days post Emergency Department
  We hypothesize that subjects managed with active rehabilitation post an acute concussion will have a 20% decreased relative risk of PCS compared to those managed with standard care.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
For the study, researchers will collect the age, gender, past medical history and through surveys, past, present and future symptoms after a head injury. This information will be used to determine which age groups are at risk and which constellation of symptoms persist following an acute head injury. All research documents and PHI will be kept in a locked cabinet and a password protected RedCap database that only study staff personnel have access to. No data will be shared until manuscript is written, but will only be shared in manuscript and not in individual data. If significant adverse data is found for a patient, the Lead PI will discuss with the subject and primary care physician.